CLINICAL TRIAL: NCT02547415
Title: Study of Characteristics of Medically Unexplained Chronic Pain in Children and Adolescents.
Brief Title: Chronic Pain in Children and Adolescents.
Acronym: PEDOUL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1408152; 2014-A01384-43 (Other: ANSM)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pain, Chronic
Keywords: Pain, Chronic; children
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires; Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with questionnaires and psychological testing: children and adolescents with chronic pain without proven medical cause, type painful somatic complaints
  Interventions: Other: questionnaires and psychological testing

INTERVENTIONS:
Other: questionnaires and psychological testing — Child/adolescent and parents interview and consultation with both a physician and a psychologist for a somatic and pain indicators assessment within an usual setting.
  Then, parents and child or adolescent are interviewed separately using different psychological instruments with only a psychologist:
  * Psychological (cognitive and projective evaluation) : Intellectual Quotient, mental flexibility, projective evaluation with Rorschach and Thematic Apperception Test, parents and children attachment questionnaires
  * Psychopathological: anxiety and depression questionnaires, psychiatric disorders evaluation, quality of life, life events questionnaires, family functioning interview.

SUMMARY:
Medically unexplained chronic pain - without identifiable somatic origin - is yet an insufficiently known and explored field in children and adolescents by international clinical works. This research aims to characterize somatic, psychological, psychopathological and environmental (particularly attachment styles and family functioning) processes trough an observational study with three pain management centers.

The study concerns children and adolescents from 7 to 17 years old, suffering of medically unexplained chronic pain and their parents who are referred to a pain center. It is composed of a somatic, psychological and family functioning assessment on the one hand and psychopathological and attachment evaluation on the other hand.

DETAILED DESCRIPTION:
Participation in the study involves an additional visit to 1 day pain center to answer questionnaires about anxiety, family environment, depression and psychological testing

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescent with chronic pain no proven medical cause, type of painful somatic complaints within the scope of one of the following diagnoses to ICD-10 (International Classification of Diseases) and DSM-IV and DSM-V (Diagnostic and Statistical Manual of Mental Disorders) to somatoform disorders, distinguishing between :

  * pain disorder
  * somatoform disorder
  * undifferentiated somatoform disorder
* Addressed to the pain centers or in pediatric chronic pain services hosting children.
* being fluently French-speaking and French-reading

Exclusion Criteria:

presence of current or past organic pathology including migraines and epilepsy, which may interfere with somatic expression of studied disorder

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescent with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Explanatory factors for pain | 1 month
  Environmental, familial, personal factors in children with chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie PERRIN, Principal Investigator — CHU de SAINT-ETIENNE
Locations (4):
- France (4):
  - Hospices Civils de LYON, Bron
  - Hopital TROUSSEAU, Paris
  - Hopital NECKER, Paris
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No